CLINICAL TRIAL: NCT04911023
Title: Comparison of Fissurectomy to Fissurectomy With Anoplasty
Acronym: ANOFIS
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ANOFIS
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Fissure Rectal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients operated by fissurectomy
- Patients operated by fissurectomy with anoplasty

SUMMARY:
Surgery is sometimes necessary to relieve patients with chronic anal fissure. It consists of resecting the edges of the fissure to make a wound larger than the initial fissure, in order to obtain healing. Thus, the edges of the wound do not stick together and the healing is done from the bottom of the wound. This procedure is widely performed in France with results that seem satisfactory. In addition to resection of the fissure, a partial closure of the wound can be associated with a small flap of rectal mucosa which is sutured with a few absorbable stitches: this is anoplasty.

DETAILED DESCRIPTION:
There is some debate as to whether to perform a fissurectomy alone or to complement it with an anoplasty to accelerate healing. The choice of technique performed depends on the training and habits of the operators but the results of fissurectomy alone and fissurectomy with anoplasty have never been compared. In the medical-surgical proctology department of the Groupe Hospitalier Paris Saint-Joseph (GHPSJ), both procedures are performed. The investigators therefore decided to compare the after-effects of fissurectomies alone with those of fissurectomies with anoplasty that were performed in the department in 2019. The choice between the 2 procedures is left exclusively to the discretion of the operator. The criteria for choice between the two patient populations are not different.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient managed in the proctology department of Groupe hospitalier Paris Saint-Joseph for single posterior idiopathic fissures (anoplasty possible only in the context of non-infected posterior fissure) between January 1 and December 31, 2019 by fissurectomy alone or fissurectomy with anoplasty

Exclusion Criteria:

* anterior or bipolar fissure
* infected fissure
* history of proctological surgery
* Crohn's disease
* HIV infection
* tubercular lesion validated by anatomopathology
* history of pelvic-perineal radiotherapy
* Tumor cells on histology
* fissurectomy +/- anoplasty associated with another proctological surgical procedure
* patient under guardianship or curatorship
* patient deprived of liberty
* patient under court protection
* Patient opposing the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected based on procedure coding:
  * HKFA004 = Excision of an anal fissure [Anal fissurectomy]
  * HKFA005 = Excision of a fissure and/or anal stenosis, with mucosal anoplasty
  * HKFA002 = Resection of an infected anal fissure
  * HKFA006 = Excision of an anal fissure, with mucosal anoplasty and resection of an isolated hemorrhoidal pack.
  The follow-up of the patients corresponds to the usual follow-up of the patients within the proctology unit (consultation at Day 15, Day 30 post-operative and then every month until complete healing).
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Compare the effectiveness of the two techniques on the disappearance of pain related to anal fissure | Day 15
  Difference between the 2 groups in terms of percent of patients free of pain at Day 15 postoperatively

SECONDARY OUTCOMES:
Compare the two techniques for the rate of complications | Day 15
  Difference between the 2 groups of patients at Day 15 post-operative in terms of complication rate
Compare the two techniques for the healing rate | Day 15
  Difference between the 2 groups of patients at Day 15 post-operative in terms of healing rate
Compare the two techniques for the rate of non-healing | Day 15
  Difference between the 2 groups of patients at Day 15 post-operative in terms of non-healing rate
Compare the two techniques for the recurrence rate | Day 15
  Difference between the 2 groups of patients at Day 15 post-operative in terms of revision rate
Compare the two techniques for the rate of revision surgery | Day 15
  Difference between the 2 groups of patients at D15 postoperatively in terms of revision rate
Search for predictive factors of failure of each technique | Day 15
  Uni- and multivariate analyses to identify risk factors for failure for each technique

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Skoufou M, Lefevre JH, Fels A, Fathallah N, Benfredj P, de Parades V. Fissurectomy with mucosal advancement flap anoplasty: The end of a dogma? J Visc Surg. 2023 Oct;160(5):330-336. doi: 10.1016/j.jviscsurg.2023.03.003. Epub 2023 Mar 25. PMID 36973105